CLINICAL TRIAL: NCT00982163
Title: A Single-Center Evaluation of the Pattern of Allergic Signs and Symptoms During 4 Weeks in Ragweed Season
Status: Completed | Type: Observational
Sponsor: ORA, Inc. (Industry)
Responsible Party: Paul Gomes, Ophthalmic Research Associates
Other Study IDs: 08-003-26
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study was designed to evaluate the pattern of seasonal allergic signs and symptoms consistent with ongoing ocular allergic inflammation during ragweed season. It was hypothesized that a pattern of ongoing ocular allergic inflammation existed in certain subjects.

DETAILED DESCRIPTION:
Subjects who had a positive skin test to ragweed within 24 months of Visit 1 were instructed to complete a diary, which assessed their allergic signs and symptoms 3 times a day for 4 weeks. During the in-office visits, subjects were asked to completed a quality of life questionnaire, as well as a retrospective and/or prospective eye allergy questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must:

  1. be willing and able to read, sign, and date the informed consent and HIPAA documents prior to initiation of Visit 1 procedures or exams;
  2. be at least 18 years of age;
  3. be willing to avoid disallowed medication, such as anti-allergy therapies
  4. have a positive history of ocular allergies and a positive skin test reaction to ragweed within the past 24 months;
  5. have a calculated logMAR visual acuity score using the ETDRS Chart of 0.60 or better in each eye at Visit 1;

Exclusion Criteria:

* Subjects may not:

  1. have preauricular lymphadenopathy or any ocular condition that could affect study parameters (particularly, clinically significant blepharitis, follicular conjunctivitis and iritis);
  2. have had any ocular infection within the last 30 days;
  3. have a positive diagnosis of moderate to severe dry eye syndrome (i.e., requiring daily use of artificial tears);
  4. wear contact lenses to each office visit; Note: Subjects will be allowed to use cold compresses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A community sample of subjects with allergic conjunctivitis and at least 18 years of age were enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Diary Data | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: H. Jerome Crampton, M.D., Principal Investigator — ORA, Inc.
Locations (1):
- ORA, Inc., North Andover, Massachusetts, United States